CLINICAL TRIAL: NCT04848857
Title: The Efficacy and Safety of Colchicine in Improving the Stability of Coronary Plaque in Patients With Acute Coronary Syndrome
Brief Title: Colchicine for the Stability of Coronary Plaque in Acute Coronary Syndrome (COLOCT)
Acronym: COLOCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, professor, director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTACS202001
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): colchicine (0.5mg), one pill a day, oral intake
  Interventions: Drug: Colchicine
- Control Group (Placebo Comparator): placebo, one pill a day, oral intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — colchicine is a potent anti-inflammatory drug which is currently recommended for the treatment of pericarditis and acute gout attacks, but also familial Mediterranean fever and Behçet disease. This drug acts on inflammation through inhibition of microtubule polymerization by binding free tubule dimers. Colchicine blunts monocyte and neutrophil invasion at the site of inflammation and reduces intracellular trafficking and thus the release of cytokine and production of reactive oxygen species and a variety of proteolytic enzymes.
  Arms: Treatment Group
Drug: Placebo — the placebo is a drug with no chemical effects but with the same physical characteristics as the experiment drug colchine.
  Arms: Control Group

SUMMARY:
Evidence from the COLCOT Trial has shown that anti-inflammatory effect of colchicine reduced the risk of cardiovascular events in patients with recent myocardial infarction. We hypothesized that this might be due to the improvement of the coronary plaque stability by colchicine. Optical coherence tomography (OCT) is the most precise method to detect plaque stability in clinical practice. Thus, the purpose of this study is to evaluate the efficacy and safety of colchicine on improving the stability of coronary plaque in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled clinical trial. OCT coronary images analyzed at an independent imaging core laboratory (Department of Cardiology, Second Affiliated Hospital of Harbin Medical University, Harbin, China) by blinded expert readers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand and sign the informed consent form voluntarily.
2. Age ≥ 18 years old and ≤ 80 years old, regardless of sex.
3. hospitalized patients diagnosed with acute coronary syndrome within 1 month.
4. at least one non-culprit lesion with diameter stenosis percentage of 30% to 70% by visual estimation on coronary angiography (CAG) after completing any planned percutaneous revascularization.
5. the lesion shown by OCT was lipid-rich plaque (Lipid pool arc > 90 °).

Exclusion Criteria:

1. Allergic to colchicine.
2. Colchicine was taken within 10 days before randomization.
3. Abnormal liver function (ALT > 3 times the upper limit of normal value).
4. Abnormal renal function (creatinine clearance rate < 45 ml/min).
5. Thrombocytopenia (PLT < 100G/L).
6. Uncontrolled infectious diseases during the screening period.
7. Known immune diseases or immune-related diseases such as systemic lupus erythematosus, asthma, inflammatory bowel disease, gout, malignant tumor and so on.
8. Pre-existing or plan for the administration of systemic anti-inflammatory treatments such as non-steroidal anti-inflammatory drugs, hormones, immunomodulatory and chemotherapeutic drugs.
9. History of surgery or interventional therapy within 6 months prior to the screening period.
10. A history of coronary artery bypass grafting or a plan for coronary artery bypass grafting within 1 year.
11. Left main coronary disease (≥50% reduction in lumen diameter by angiographic visual estimation).
12. Significant coronary calcification or tortuosity deemed to preclude OCT evaluation.
13. Diagnosed with mental disorders such as anxiety or depression.
14. Pregnant women, lactating women or women of childbearing age who do not use effective contraceptive methods.
15. Participated in other clinical trials within 3 months before the screening period.
16. Do not receive standardized treatment after being diagnosed with coronary heart disease.
17. The life expectancy of the subjects is less than 1 year.
18. The researchers determined that other conditions in which the patient was not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
changes of the Thickness of fibrous cap of coronary artery plaque | 12 months
  changes of the thickness of fibrous cap of coronary artery plaque measured by OCT

SECONDARY OUTCOMES:
changes of the Average lipid arc of coronary artery plaque | 12 months
  changes of the average lipid arc of coronary artery plaque measured by OCT
changes of the Macrophage accumulation in coronary artery plaque | 12 months
  changes of the macrophage accumulation in coronary artery plaque measured by OCT
changes of the Incidence of thin-cap fibroatheroma (TCFA) | 12 months
  changes of the incidence of TCFA measured by OCT
changes of the Minimum lumen area (MLA) | 12 months
  changes of the MLA measured by OCT
changes of the inflammatory biomarkers (hsCRP, IL-6, and MPO) | 12 months
  changes of the inflammatory biomarkers (hsCRP, IL-6, and MPO)
major adverse cardiovascular and cerebrovascular events (MACCEs) | 12 months
  A composite of all-cause death, nonfatal myocardial infarction, nonfatal stroke, revascularization due to ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yu M, Yang Y, Dong SL, Zhao C, Yang F, Yuan YF, Liao YH, He SL, Liu K, Wei F, Jia HB, Yu B, Cheng X. Effect of Colchicine on Coronary Plaque Stability in Acute Coronary Syndrome as Assessed by Optical Coherence Tomography: The COLOCT Randomized Clinical Trial. Circulation. 2024 Sep 24;150(13):981-993. doi: 10.1161/CIRCULATIONAHA.124.069808. Epub 2024 Aug 21. PMID 39166327